CLINICAL TRIAL: NCT04246229
Title: Transcutaneous Bilirubinometry in Neonatal Hyperbilirubinemia During and After Phototherapy: a Randomized Controlled Trial
Brief Title: Transcutaneous Bilirubinometry and Phototherapy
Acronym: TRABIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Principal Investigator, Jolita Bekhof, MD PhD Principal Investigator, Princess Amalia Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 202001
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: transcutaneous bilirubinometry; phototherapy; neonatal icterus; neonatal jaundice; newborn
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous bilirubinometry (Experimental): in this arm the bilirubin level to monitor the effect of phototherapy will be measured through transcutaneous mbiirubinometry
  Interventions: Diagnostic Test: Transcutaneous bilirubinometry
- serum bilirubin (Active Comparator): In this arm the bilirubin level to monitor the effect of phototherapy wil be measured through measurements of serum bilirubin obtained through blood draws
  Interventions: Diagnostic Test: Serum bilirubin

INTERVENTIONS:
Diagnostic Test: Transcutaneous bilirubinometry — use of transcutaneous bilirubinometry a non-invasieve measurement of skin bilirubin levels
  Arms: transcutaneous bilirubinometry
Diagnostic Test: Serum bilirubin — use of blood draws to measure serum bilirubin level
  Other Names: blood draw
  Arms: serum bilirubin

SUMMARY:
A randomized Controlled trial comparing the use of transcutaneous bilirubinometry to serum bilirubin measurements (via blooddraws = standard care) in neonates born after a gestational age > 32 weeks and < 15 days of age treated with Phototherapy for neonatal hyperbilrubinemia.

DETAILED DESCRIPTION:
A randomized Controlled trial comparing the use of transcutaneous bilirubinometry to serum bilirubin measurements (via blooddraws = standard care) in neonates born after a gestational age > 32 weeks and < 15 days of age treated with Phototherapy for neonatal hyperbilrubinemia. Main outcome measurement is the number of blooddraws for measurement of bilirubin. Secondary outcome measurements are duration of phototherapy and hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with indication for phototherapy for treatment of hyperbilirubinemia

Exclusion Criteria:

* skinlesions located on the sternum interfering with transcutaneous measurement
* exchange transfusion

Ages: 0 Days to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
blood draws | during hospitalisation with a maximum of 14 days
  number of blood draws from the start of phototherapy for measurement of serum bilirubin

SECONDARY OUTCOMES:
phototherapy duration | during hospitalisation with a maximum of 14 days
  duration of phototherapy in hours
hospitalisation | 3 months
  duration of hospitalisation in days

CONTACTS AND LOCATIONS:
Overall Officials: Jolita Bekhof, MD,PhD, Principal Investigator — 1971
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After publishing the results the individual participant data will be anonimously available upon request
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after publication in a peer reviewed journal during 3 years
Access Criteria: relevant research question